CLINICAL TRIAL: NCT05443477
Title: To Evaluate the Improvement Effect of Supplementing Hericium Erinaceus Mycelium Capsules and Grape King Probiotic Capsules of the Grape King Bio on Physiological and Psychological Symptoms of Premenstrual Syndrome
Brief Title: Hericium Erinaceus Mycelium and Probiotic of the Grape King Bio on Symptoms of Premenstrual Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CS2-20104; BR-CT004 (Other Grant/Funding Number: Grape King Bio)
Record Dates: First submitted 2022-06-12; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Hericium Erinaceus mycelium; probiotic
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: In the intervention phase of this study, 105 eligible participant were randomly divided into intervention (Grape King Hericium erinaceus Mycelium Capsules and Grape King Probiotic Capsules) and placebo groups (n=35/group). Both subjects and researchers were blind to the treatment assignment until the statistical analysis was completed.
Who Masked: Participant, Investigator
Masking Description: Both subjects and researchers were blind to the treatment assignment until the statistical analysis was completed. All the subjects were randomly divided into placebo group and two intervention groups (i.e. supplementation with Grape King Hericium erinaceus Mycelium Capsules and Grape King Probiotic Capsules) by using Excel to generate random numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hericium Erinaceus Mycelium (Experimental): patients with premenstrual syndrome received supplementation of Hericium Erinaceus Mycelium capsules
  Interventions: Dietary Supplement: Hericium Erinaceus Mycelium
- Probiotic (Experimental): patients with premenstrual syndrome received supplementation of Probiotic capsules
  Interventions: Dietary Supplement: Probiotic
- control (Placebo Comparator): patients with premenstrual syndrome received supplementation of placebo capsules
  Interventions: Dietary Supplement: control

INTERVENTIONS:
Dietary Supplement: Hericium Erinaceus Mycelium — participants received two oral capsules containing Hericium erinaceus Mycelium every day for the 3 months.
  Arms: Hericium Erinaceus Mycelium
Dietary Supplement: Probiotic — participants received two oral capsules containing Probiotic powder every day for the 3 months.
  Arms: Probiotic
Dietary Supplement: control — participants received two oral capsules containing control powder every day for the 3 months.
  Arms: control

SUMMARY:
The purpose of this experiment is to evaluate the efficacy of supplemental health food Grape King Hericium erinaceus Mycelium Capsules and Grape King Probiotic Capsules in improving physical and psychological symptoms, blood oxidative stress and inflammation indicators in women with premenstrual syndrome.

DETAILED DESCRIPTION:
This study was a randomized, double-blinded and placebo-controlled research. This study was approved by the Institutional Review Board of the Chung Shan Medical University Hospital and all Participants signed the written informed consent to participate in the study.

Participants met the inclusion criteria, ie: age 20~45 yr and a regular menstrual cycle (21~35 days per cycle) were recruited through advertisements posted around the Chun Shan Medical university campus. In screening phase of this study, affective and one somatic symptom in before onset of menstruation in two consecutive cycles and was not affected by depression or anxiety disorder, she is examined by the Attending Physician of the Obstetrics and Gynecology Department to diagnosed a patient with premenstrual syndrome. In the intervention phase of this study, 105 eligible participant were randomly divided into intervention (Grape King Hericium erinaceus Mycelium Capsules and Grape King Probiotic Capsules) and control groups (n=35/group). Both subjects and researchers were blind to the treatment assignment until the statistical analysis was completed. All participants received two oral capsules containing Hericium erinaceus Mycelium, probiotics or placebo every day for the 3 months. The capsules of intervention supplementations and placebo provided by Grape King Biotechnology Inc in identical appearance and package to guarantee the blindness.

Data collection A validated semi-quantitative Food Frequency Questionnaire was used to obtain daily nutritional values of participants. To assess the symptoms of PMS, all subjects need to fill out daily record of severity of problems on a daily basis in the 3 months of intervention period and 6 months after the intervention. In the 0, 1, 3 months of intervention, the anthropometric parameters and body composition were measured by using bioelectrical impedance analysis method ( MC-980 MA PLUS, TANITA BIA Technology). In the 0, 1, 3 months of intervention, venous blood samples were taken from all subjects for measuring the marks of oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-45
2. The menstrual cycle is 21~35 days/time
3. PMS diagnosed by an obstetrician
4. Willing to sign the subject's consent form

Exclusion Criteria:

1. Those are with cancer, cardiovascular, kidney, liver, infectious and endocrine diseases, aw well as with depression and anxiety tendencies
2. Those have a surgery in the last 6 months
3. Those use of probiotics, estrogen and birth control pills
4. Body mass index > 39 kg/m2, smoking, drinking
5. Death of a close relative and other stressful events within the last 6 months

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women who are menstruating
Enrollment: 105 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-01-07 (Estimated); Study Completion 2023-01-07 (Estimated)

PRIMARY OUTCOMES:
The differences from control of Daily record of severity of problems | All eligible subjects recorded their symptoms by questionnaire of daily record of severity of problems at every day of 3 consecutive menstrual cycles during the intervention period and the 3rd menstrual cycles at the end of intervention.
  This questionnaire of daily record of severity of problems were using to determine the severity of PMS including mood, physical and behavioral symptoms and characteristics. There are21 items grouped into 11 domains. Additional questions asked about quality of life and satisfaction of self-health. The levels of severity on this form are: 1- Not at all, 2- Minimal to Mild, 3-Moderate, 4- Severe. During each month of the intervention period and the 3rd menstrual cycles at the end of intervention, the differences of the total scores of menstrual cycles compared with the control group in each intervention groups were analyzed.
The changes from baseline of Daily record of severity of problems | All eligible subjects recorded their symptoms by questionnaire of daily record of severity of problems at every day of 3 consecutive menstrual cycles during the intervention period and the 3rd menstrual cycles at the end of intervention.
  This questionnaire of daily record of severity of problems were using to determine the severity of PMS including mood, physical and behavioral symptoms and characteristics. There are21 items grouped into 11 domains. Additional questions asked about quality of life and satisfaction of self-health. The levels of severity on this form are: 1- Not at all, 2- Minimal to Mild, 3-Moderate, 4- Severe. During each month of the intervention period and the 3rd menstrual cycles at the end of intervention, the changes of the total scores of menstrual cycles compared with the baseline in each groups were analyzed.

SECONDARY OUTCOMES:
The differences from control of high-sensitivity C-reactive protein | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of high-sensitivity C-reactive protein.
  The inflammation marker, high-sensitivity C-reactive protein (mg/L), in the blood of the subjects were measured. The different concentration of the high-sensitivity C-reactive protein at each time points of intervention groups compared with control group were analyzed.
The differences from baseline of high-sensitivity C-reactive protein | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of high-sensitivity C-reactive protein.
  The inflammation marker, high-sensitivity C-reactive protein (mg/L), in the blood of the subjects were measured. The different concentration of the high-sensitivity C-reactive proteinat at the 1st and 3rd month compared with baseline in each group were analyzed.
The differences from control of high-sensitivity interleukin-6 | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of interleukin-6.
  The inflammation marker, interleukin-6 (pg/mL), in the blood of the subjects were measured. The different concentration of the interleukin-6 at each time points of intervention groups compared with control group were analyzed.
The differences from baseline of high-sensitivity interleukin-6 | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of interleukin-6.
  The inflammation marker, interleukin-6 (pg/mL), in the blood of the subjects were measured. The different concentration of the interleukin-6 at the 1st and 3rd month compared with baseline in each group were analyzed.
The differences from control of high-sensitivity interleukin-1 | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of interleukin-1.
  The inflammation marker, interleukin-1 (pg/mL), in the blood of the subjects were measured. The different concentration of the interleukin-1 at each time points of intervention groups compared with control group were analyzed.
The differences from baseline of high-sensitivity interleukin-1 | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of interleukin-1.
  The inflammation marker, interleukin-1 (pg/mL), in the blood of the subjects were measured. The different concentration of the interleukin-1 at the 1st and 3rd month compared with baseline in each group were analyzed.
The differences from control of high-sensitivity TNF-a | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of TNF-a.
  The inflammation marker, TNF-a (pg/mL), in the blood of the subjects were measured. The different concentration of the TNF-a at each time points of intervention groups compared with control group were analyzed.
The differences from baseline of high-sensitivity TNF-a | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of TNF-a.
  The inflammation marker, TNF-a (pg/mL), in the blood of the subjects were measured. The different concentration of the TNF-a at the 1st and 3rd month compared with baseline in each group were analyzed.
The differences from control of total antioxidant capacity | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of total antioxidant capacity.
  The oxidative stress index, total antioxidant capacity (μmol/L), in the blood of the subjects were measured. The different concentration of the total antioxidant capacity at each time points of intervention groups compared with control group were analyzed.
The differences from baseline of total antioxidant capacity | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of total antioxidant capacity.
  The oxidative stress index, total antioxidant capacity (μmol/L), in the blood of the subjects were measured. The different concentration of the total antioxidant capacity at the 1st and 3rd month compared with baseline in each group were analyzed.
The differences from control of malondialdehyde | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of malondialdehyde.
  The oxidative stress index, malondialdehyde (nmol/mL), in the blood of the subjects were measured. The different concentration of the total antioxidant capacity at each time points of intervention groups compared with control group were analyzed.
The differences from baseline of malondialdehyde | In the 1st data of menstruation of the beginning, 1st and 3rd months of intervention, the blood of all eligible subjects were collected to measure the concentration of malondialdehyde.
  The oxidative stress index, malondialdehyde (nmol/mL), in the blood of the subjects were measured. The different concentration of the total antioxidant capacity at the 1st and 3rd month compared with baseline in each group were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Li Liu, PhD, Study Chair — Department of Nutrition, Chung Shan Medical University, Taichung, Taiwan; Man-Jung Hung, MD, PhD, Principal Investigator — Department of Medicine, Chung Shan Medical University, Taichung, Taiwan; Yi-Chin Lin, PhD, Principal Investigator — Department of Nutrition, Chung Shan Medical University, Taichung, Taiwan; Pey-Ling Shieh Shieh, PhD, Principal Investigator — Department of Psychology, Chung Shan Medical University, Taichung, Taiwan
Locations (1):
- Kai-Li Liu, Taichung, Taiwan

REFERENCES:
- [Result] Duvan CI, Cumaoglu A, Turhan NO, Karasu C, Kafali H. Oxidant/antioxidant status in premenstrual syndrome. Arch Gynecol Obstet. 2011 Feb;283(2):299-304. doi: 10.1007/s00404-009-1347-y. Epub 2010 Jan 19. PMID 20084389
- [Result] Danis P, Drew A, Lingow S, Kurz S. Evidence-based tools for premenstrual disorders. J Fam Pract. 2020 Jan/Feb;69(1):E9-E17. No abstract available. PMID 32017837
- [Result] Endicott J, Nee J, Harrison W. Daily Record of Severity of Problems (DRSP): reliability and validity. Arch Womens Ment Health. 2006 Jan;9(1):41-9. doi: 10.1007/s00737-005-0103-y. Epub 2005 Sep 20. PMID 16172836
- [Result] Sharifi-Rad J, Rodrigues CF, Stojanovic-Radic Z, Dimitrijevic M, Aleksic A, Neffe-Skocinska K, Zielinska D, Kolozyn-Krajewska D, Salehi B, Milton Prabu S, Schutz F, Docea AO, Martins N, Calina D. Probiotics: Versatile Bioactive Components in Promoting Human Health. Medicina (Kaunas). 2020 Aug 27;56(9):433. doi: 10.3390/medicina56090433. PMID 32867260
- [Result] Nagano M, Shimizu K, Kondo R, Hayashi C, Sato D, Kitagawa K, Ohnuki K. Reduction of depression and anxiety by 4 weeks Hericium erinaceus intake. Biomed Res. 2010 Aug;31(4):231-7. doi: 10.2220/biomedres.31.231. PMID 20834180